CLINICAL TRIAL: NCT02417753
Title: A Pilot Study of AZD9150, a STAT3 Antisense Oligonucleotide in Malignant Ascites
Brief Title: AZD9150, a STAT3 Antisense Oligonucleotide, in People With Malignant Ascites
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed because we could not find these types of patients.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., National Cancer Institute, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150112; 15-C-0112
Record Dates: First submitted 2015-04-15; First posted 2015-04-16 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms; Ascites; Gastrointestinal Cancer; Gastrointestinal Neoplasms
Keywords: PARACENTESIS; STAT3 Antisense Oligonucleotide; Ascites; AZD9150; Surgical Resection
MeSH Terms: conditions — Ovarian Neoplasms; Ascites; Gastrointestinal Neoplasms | interventions — danvatirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD9150 in People with Malignant Ascites (Experimental): AZD9150 over a 28 day cycle
  Interventions: Drug: AZD9150

INTERVENTIONS:
Drug: AZD9150 — AZD9150 IV infusion over 3 hours Cycle 1: days 1, 3, 5, 8, 15 and 22 of a 28 day cycle. Cycle 2 and beyond Days 1, 8, 15 and 22 of a 28 day cycle

SUMMARY:
Background:

- Some people with gastrointestinal or ovarian cancer also have ascites. That is free fluid built up in the abdomen. Researchers want to see if a new drug can affect some of the immune cells in the ascites. This may also treat the cancer.

Objective:

- To look at the immune markers the ascites of people with gastrointestinal or ovarian cancer.

Eligibility:

- Adults age 18 and older with a malignancy of the gastrointestinal tract (GI) tract or metastatic ovarian cancer. As a result, they have ascites in the abdomen.

Design:

* Participants will be screened with:
* Medical history, physical exam, and blood tests.
* Echocardiogram: sound waves make images of the heart.
* Electrocardiogram: measures electrical activity of the heart.
* Paracentesis: a needle will be inserted in the abdomen and will remove some of the ascites fluid.
* They may have a tumor biopsy.
* Participants will get AZD9150 through a vein for 3 hours. They will get this 6 times in cycle 1 and 4 times all other cycles. Each cycle is 28 days.
* Each cycle, participants will:
* Have a physical exam.
* Have blood tests weekly.
* Be asked about how they feel and any medicines they are taking.
* After every 2 cycles (about every 2 months), participants will have scans and x-rays of their tumor.
* Participants will have paracentesis 2 more times during the study. They will have another echocardiogram.
* At the end of therapy, participants will have a physical exam and blood tests. They will be asked about how they feel and any medicines they are taking.

DETAILED DESCRIPTION:
Background:

* Signal transducer and activator of transcription 3 (STAT)3 is considered to be a promising cancer drug target because of its pleiotropic involvement in tumorigenesis. STAT3 not only regulates the expression of many genes which are directly important for the survival of tumor cells, but it is also an important factor in non-tumor cells in the tumor microenvironment involved in immune evasion of tumor cells, angiogenesis, and metastasis.
* AZD9150 is an antisense oligonucleotide designed to target and down-regulate expression of human STAT3 mRNA.
* By focusing on patients with malignant ascites it will be more feasible for us to sample the tumor environment and to do it more frequently than, for example, conventional tumor tissue biopsies. Malignant ascites is a relatively common occurrence in ovarian and gastrointestinal malignancies, impacting greatly on quality of life.

Objectives:

-To measure changes in immune parameters in the malignant ascites of patients with advanced cancer following therapy with AZD9150.

Select Eligibility:

* Age greater than or equal to 18 years.
* Histologically confirmed metastatic ovarian or GI malignancy with malignant ascites. Patients must have ascites amenable for paracentesis.
* Patient that have relapsed or have been refractory to at least one prior chemotherapy regimen, or patients for whom no standard therapy exists

Design:

* Up to N=15 eligible patients will receive AZD9150 at the following schedule:

  * Cycle 1 only: AZD9150 will be administered intravenously on Cycle 1 Days 1, 3, 5, 8, 15 and 22.
  * Cycle 2 and beyond: AZD9150 will be administered as an intravenous infusion every week without break, i.e. Days 1, 8, 15 and 22 of a 28-day cycle.
* Patients will be re-staged every 8 weeks.
* Patients will undergo a baseline pretreatment paracentesis which will be repeated on Cycle 1 Days 8 and 15. An optional paracentesis may be attempted on D57 or off treatment (whichever happens first). Immune subsets analysis at baseline in biopsy/ascites/peripheral blood mononuclear cells (PBMC) and post AZD9150 in surgical specimen, ascites and PBMC will be analyzed. STAT3 activation status will also be assessed in tumor cells isolated from malignant ascites at various time points.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have histologically or cytologically confirmed gastrointestinal (G)I malignancies or ovarian cancer prior to entering this study.
2. Histologically confirmed metastatic ovarian or GI malignancy with malignant ascites amenable for paracentesis. Adjudication of malignant ascites can be made on clinical grounds e.g. in the absence of cirrhosis or other non-malignant causes of ascites.
3. Patients who have relapsed or are refractory to at least one prior chemotherapy regimen, and for whom no standard therapy exists. There is no limit to the number of prior chemotherapy regimens received.
4. Patients should be off radiation therapy, chemotherapy, investigational agents, hormonal therapy, or immunotherapy for 4 weeks (or 5 half-lives of the therapy, whichever is longer) prior to first dose in the study, and off Bevacizumab 6 weeks.
5. Age greater than or equal to 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >70%)
7. Patients must have normal organ and marrow function as defined below:

   * leukocytes >3,000/mcL
   * absolute neutrophil count >1,500/mcL without growth-factor support during the past month
   * platelets >100,000/mcL at all times during the screening period without platelet transfusion within 3 weeks

     -total bilirubin <2 X institutional upper limit of normal
   * Hemoglobin (Hb) greater than or equal to 9 g/dL without transfusion for 3 weeks
   * International normalized ratio (INR) < 2.0
   * Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase (SGPT) <3 X institutional upper limit of normal, or <5 ULN for patients with liver metastasis
   * Creatinine within normal institutional limits

   OR
8. Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be < grade 1
9. Ejection fraction > 50% on echocardiogram.
10. The effects of AZD9150 on the developing human fetus are unknown. For this reason women of child-bearing potential should use reliable methods of contraception from the time of screening until 6 months after discontinuing study treatment. Acceptable methods of contraception include tubal ligation, tricycle combined oral or transdermal contraceptives, copper-banded intra-uterine devices and vasectomized partner. It is not known whether AZD9150 has the capacity to induce hepatic enzymes so hormonal contraceptives should be combined with a barrier method of contraception. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women of child-bearing potential must have a negative pregnancy test prior to entry. Male patients should use reliable methods of contraception such as barrier contraception i.e. condoms during sexual activities with women of child-bearing potential and refrain from sperm donation during the trial and for a washout period of at least 6 months. If male patients wish to father children they should be advised to arrange for freezing of sperm samples prior to the start of study treatment.
11. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Patients who are receiving any other investigational agents.
2. History of prior Janus kinase (JAK) or signal transducer and activator transcription 3 (STAT)3 inhibitor treatment.
3. Patients with known brain metastases or spinal cord compression should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. Patients must not have other invasive malignancies within the past 3 years (with the exception of adequately treated basal or squamous cell skin cancers, carcinoma in situ of the cervix and ductal carcinoma in situ (DCIS) of breast).
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD9150.
6. Incompletely healed surgical incision prior to enrolment
7. Ongoing therapy with oral or parenteral anticoagulants (e.g., heparin, warfarin). Lowdose anticoagulants for maintenance of catheter patency are not exclusionary.
8. Any of the following cardiac criteria:

   * Mean resting corrected Q wave and T wave (QT) interval (QTcF) > 480 msec obtained from 3 electrocardiograms (ECGs)
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g., complete left bundle branch block, third degree heart block
9. Patients with uncontrolled hypertension (systolic blood pressure (SBP)> 155, diastolic blood pressure (DBP)> 90), unstable coronary disease (unstable angina, evidence of congestive heart failure (CHF), or myocardial infarction (MI) within 6 months of study)
10. New York Heart Association (NYHA) greater than or equal to Grade II or greater.
11. History of myocardial infarction within 6months prior to screening.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
13. Pregnant and/or breastfeeding
14. Human immunodeficiency virus (HIV)-positive patients or with history of hepatitis or with current chronic or active hepatitis. A past history of Hepatitis A is allowed.
15. History of recurrent bacterial infections unrelated to hepatocellular carcinoma (HCC) (particularly skin or lung)
16. Bacterial peritonitis within 30 days
17. History of, or presently active or chronic viral infections (i.e. zoster or hepatitis)
18. History of known latent or active tuberculosis, signs of active or latent tuberculosis on chest X-ray, skin test showing an induration of >10 mm or more or according to local recommendations.
19. Active bleeding disorders and high likelihood of bleeding or conditions or medications known to increase the risk of bleeding. Patients with bleeding diathesis and subjects who are receiving anticoagulation treatment with INR > 2 are excluded.
20. History of recurrent thrombosis or any thrombosis within the past 6 months
21. Family history consistent with thrombophilia or hypofibrinolysis
22. Patients who have received liver transplantation
23. History of clinically significant liver abnormalities other than liver metastasis
24. Presence of hepatic encephalopathy within 4 weeks of 1st dose
25. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-04-03 (Actual); Primary Completion 2016-04-07 (Actual); Study Completion 2016-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZD9150 in People With Malignant Ascites
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | AZD9150 in People With Malignant Ascites
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Changes in Immune Parameters in the Malignant Ascites of Patients With Advanced Cancer Following Therapy With AZD9150
Description: Participants were to undergo research paracentesis. Ascitic fluid was to be obtained and processed for changes in the percentages of memory cluster of differentiation 8 (CD8) + cells, regulatory T cells, plasmacytoid dendritic cell (pDC), B cells and natural killer (NK) cells will be analyzed by flow cytometry.
Time Frame: 1.5 years
Population: This outcome measure was not done because the one patient did not make it to one scan after 8 weeks.
Arm/Group | AZD9150 in People With Malignant Ascites
Number analyzed (Participants) | 0

2. Secondary Outcome: Effect on Signal Transducer and Activator of Transcription 3(STAT3)-Dependent & Associated Signaling Both in Tumor Cells, Peripheral Blood and the Microenvironment, Including Modulations in Chemokine and Cytokine Response Following Treatment With AZD9150
Description: Serum samples were to be collected from participants and assessed for interferon, cytokine and chemokine levels including interferon, ϒ-interferon inducible protein (IP-10), monocyte chemoattractant protein 1 (MCP-1), interleukin 6 (IL-6), interleukin 8 (IL-8), interleukin 10 (IL-10), and interleukin 12/p70 (IL-12/p70).
Time Frame: 1.5 years
Population: This outcome measure was not done because the one patient did not make it to one scan after 8 weeks.
Arm/Group | AZD9150 in People With Malignant Ascites
Number analyzed (Participants) | 0

3. Secondary Outcome: Reduction in Tyrosine-phosphorylated Signal Transducer and Activator of Transcription 3 (STAT3) Phospho- Signal Transducer and Activator of Transcription 3 (p- STAT3) Expression, Comparing Before and After Therapy, in Ascites and Peripheral Blood
Description: Measure the reduction in tyrosine-phosphorylated STAT3 (p=STAT3) expression.
Time Frame: 1.5 years
Population: This outcome measure was not done because the one patient did not make it to one scan after 8 weeks.
Arm/Group | AZD9150 in People With Malignant Ascites
Number analyzed (Participants) | 0

4. Secondary Outcome: Response Rate (RR) in Patients With Malignant Ascites Treated With AZD9150
Description: Response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and is measured from the time measurement criteria are met for complete response or partial response (whichever is recorded first) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: 1.5 years
Population: This outcome measure was not done because the one patient did not make it to one scan after 8 weeks.
Arm/Group | AZD9150 in People With Malignant Ascites
Number analyzed (Participants) | 0

5. Secondary Outcome: Count of Participants With Serious and Non Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 4 months and 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | AZD9150 in People With Malignant Ascites
Number analyzed (Participants) | 1
Participants | 1

6. Secondary Outcome: Progression Free Survival (PFS) in Patients With Malignant Ascites Treated With AZD9150
Description: PFS is the time interval from start of treatment to documented evidence of progressive disease. Progressive disease was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). in addition to the relative increase of 29%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 1.5 years
Population: This outcome measure was not done because the one patient did not make it to one scan after 8 weeks.
Arm/Group | AZD9150 in People With Malignant Ascites
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival (PFS) in Patients With Malignant Ascites Treated With AZD9150
Description: OS is defined as the time from the first day of treatment to the day of death.
Time Frame: 1.5 years
Population: This outcome measure was not done because the one patient did not make it to one scan after 8 weeks.
Arm/Group | AZD9150 in People With Malignant Ascites
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 months and 15 days
Arm/Group | AZD9150 in People With Malignant Ascites
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9150 in People With Malignant Ascites (N=1)
Ascites (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Edema trunk (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9150 in People With Malignant Ascites (N=1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (4)
Constipation (Gastrointestinal disorders) | 1 (3)
Creatinine increased (Investigations) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Edema limbs (General disorders) | 1 (2)
Fibrinogen decreased (Investigations) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (6)
Nausea (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No